CLINICAL TRIAL: NCT01114477
Title: NeuroStar TMS Therapy System: Data Management, Analysis and Reporting Format for Clinical Treatment Utilization and Outcomes (Protocol no. 19-50001-000,Rev D
Brief Title: NeuroStar TMS Therapy System: Utilization and Outcomes
Status: Completed | Type: Observational
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Other Study IDs: 19-50001-000
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial magnetic stimulation; TMS; Observational study; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The major objective of this observational study is to describe clinical outcomes of patients receiving treatment with the NeuroStar TMS Therapy system in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder

Exclusion Criteria:

* Contraindications to treatment with TMS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical practice locations providing clinical treatment with the NeuroStar TMS Therapy System.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Total Score on the Patient Health Questionnaire 9-Item (PHQ-9) | Baseline and 6 weeks
  The primary outcome measure will reported as the change from baseline through 6 weeks for the total score on the PHQ-9.

SECONDARY OUTCOMES:
Total score for the Clinical Global Impressions-Severity (CGI-S) | Baseline, 6 weeks and 12 Months
  The change from baseline to endpoint on the total score for the CGI-S will be reported for the 6 week and 12 month time points.
Total score for the Inventory of Depressive Symptoms-Self Report (IDS-SR) | Baseline, 6 weeks and 12 Months
  The change from baseline to endpoint on the total score for the IDS-SR will be reported for the 6 week and 12 month time points.
Total Score for the EuroQol Questionnaire (EQ-5D) | Baseline, 6 weeks, and 12 Months.
  The change from baseline to endpoint on the total score for the EQ-5D will be reported for the 6 week and 12 month time points.
Health Resource Utilization Questionnaire (HRU) | Baseline, 6 weeks, and 12 Months
  The change from baseline in health care service utilization reported on the individual questions contained in the HRU will be reported for the 6 week and 12 month time points.
Short Form 36-Item Questionnaire(SF-36) Individual Factor Scores and General Medical and Mental Health Composite Scores | Baseline, 6 weeks, and 12 Months.
  The change from baseline to endpoint on the Individual Factor Scores and General Medical and Mental Health Composite Scores for the SF-36 will be reported for the 6 week and 12 month time points.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Demitrack, MD, Study Director — Neuronetics, Inc.
Locations (44):
- United States (44):
  - Lee Ann Kelley, M.D., PC, Phoenix, Arizona
  - Bay Psychiatric Associates, Berkeley, California
  - TMS Center of Beverly Hills, Beverly Hills, California
  - Clinical Training & Research Institute, Burlingame, California
  - Sacramento TMS, El Dorado Hills, California
  - Martha Koo, MD, Hermosa Beach, California
  - Orange County TMS Center, Laguna Hills, California
  - Depression Research Center and Clinic-Semel Institute for Neuroscience & Human Behavior at UCLA, Los Angeles, California
  - Kevin Kinback, MD, Mission Viejo, California
  - Todd Hutton, MD & Associates, Pasadena, California
  - The Botkiss Center for TMS Therapy, San Diego, California
  - Stanford Hospital and Clinics, Stanford, California
  - Arjun Reyes, MD, Woodland Hills, California
  - Hartford Hospital, Hartford, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Christiana Care Health Services, Wilmington, Delaware
  - Health Sciences America, LLC, Boca Raton, Florida
  - Curtis Cassidy, MD, Lakeland, Florida
  - Brian Teliho, MD, Atlanta, Georgia
  - Carl M. Wahlstrom, Jr. MD Limited, Chicago, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Brain Stimulation Chicago North Shore, Northbrook, Illinois
  - Behavioral Health Care Associates, Schaumburg, Illinois
  - University Psychiatric Foundation, Louisville, Kentucky
  - Integrative Psychiatry, Louisville, Kentucky
  - Spectrum Behavioral Health, Annapolis, Maryland
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Anthony Drobnick, MD, Saint Michaels, Maryland
  - Newton-Wellesley Psychiatry, Newton, Massachusetts
  - Central Psychiatry, Las Vegas, Nevada
  - TMS Center of New England, Portsmouth, New Hampshire
  - Santa Fe TMS Therapy Center, Santa Fe, New Mexico
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - The TMS Institute of Pennsylvania-Advanced Neuropsychiatric Solutions, West Chester, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - W. Scott West, M.D., Nashville, Tennessee
  - Texas Neuropsychiatric Institute, Amarillo, Texas
  - Texas TMS Center at Senior Adults Specialty Healthcare (SASH), Austin, Texas
  - Houston TMS, Houston, Texas
  - Agape Mind Services/The Costello Clinic, Lewisville, Texas
  - Serenity Center for Depression, P.A., Sugar Land, Texas
  - University Neuropsychiatric Institute, Salt Lake City, Utah
  - Center for Anxiety and Depression, Mercer Island, Washington

REFERENCES:
- [Derived] Dunner DL, Aaronson ST, Sackeim HA, Janicak PG, Carpenter LL, Boyadjis T, Brock DG, Bonneh-Barkay D, Cook IA, Lanocha K, Solvason HB, Demitrack MA. A multisite, naturalistic, observational study of transcranial magnetic stimulation for patients with pharmacoresistant major depressive disorder: durability of benefit over a 1-year follow-up period. J Clin Psychiatry. 2014 Dec;75(12):1394-401. doi: 10.4088/JCP.13m08977. PMID 25271871
- [Derived] Janicak PG, Dunner DL, Aaronson ST, Carpenter LL, Boyadjis TA, Brock DG, Cook IA, Lanocha K, Solvason HB, Bonneh-Barkay D, Demitrack MA. Transcranial magnetic stimulation (TMS) for major depression: a multisite, naturalistic, observational study of quality of life outcome measures in clinical practice. CNS Spectr. 2013 Dec;18(6):322-32. doi: 10.1017/S1092852913000357. Epub 2013 Jul 30. PMID 23895940